CLINICAL TRIAL: NCT06532396
Title: A Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of QRL-101 in Healthy Participants
Brief Title: A Study Evaluating Multiple Ascending Doses of QRL-101 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-101-03
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; QRL-101

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, double-blind, placebo-controlled multiple ascending dose (MAD) study in healthy participants with the primary goal of evaluating the safety and tolerability of QRL-101.
Who Masked: Participant, Investigator
Masking Description: A participant and investigator-blinded, randomized, placebo-controlled design will be used to minimize bias in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QRL-101 (Experimental): Multiple-ascending doses of QRL-101 will be administered orally to healthy participants.
  Interventions: Drug: QRL-101
- Placebo (Placebo Comparator): Multiple-ascending doses of comparator placebo will be administered orally to healthy participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QRL-101 — Multiple-ascending doses of QRL-101 will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Arms: QRL-101
Drug: Placebo — Multiple-ascending doses of comparator placebo will be administered orally to healthy participants.
  Arms: Placebo

SUMMARY:
QRL-101-03 is a multiple ascending dose (MAD) study to evaluate the safety, tolerability, and pharmacokinetics (PK) of QRL-101 in healthy participants. QRL-101-03 is a follow-on study to QRL-101-01, an ongoing Phase 1, single ascending dose study to determine the safety, tolerability, and PK profile of QRL-101 after a single dose (ClinicalTrials.gov ID: NCT05667779).

DETAILED DESCRIPTION:
Phase 1, single-site, multiple-dose study to evaluate the safety, tolerability, and PK of multiple ascending doses of QRL-101 in healthy participants. Up to 5 cohorts of 8 participants each, randomized 6:2 (QRL-101: placebo) will be tested. The approximate total duration of study participation for each participant may be up to 39 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years of age inclusive at the time of signing the informed consent.
2. Clinical chemistry laboratory values within acceptable range for the population, as per investigator judgment.
3. Body mass index of 18 to 32 kg/m2 (inclusive).
4. Willing and able to practice effective contraception.

Exclusion Criteria:

1. Currently enrolled in any other clinical trial involving a study drug or off-label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Any participant in >4 studies a year and/or has participated in a clinical trial within 1 month of expected dosing date.
3. History or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more treatment emergent adverse events and serious adverse events. | Baseline through Follow up (Day 10)
  A summary of treatment emergent adverse events (AEs), serious adverse events (SAEs), and other non-serious adverse events, regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Pharmacokinetics (plasma): Area under the concentration time curve during the dosing interval (AUCτ) of QRL-101 | Baseline through Follow up Day 5
  Area under the concentration time curve during the dosing interval (AUCτ) of QRL-101
Pharmacokinetics (plasma): Maximum observed concentration of QRL-101 | Baseline through Follow up Day 5
  Maximum observed concentration (Cmax) of QRL-101
Pharmacokinetics (plasma): Time of maximum concentration of QRL-101 | Baseline through Follow up Day 5
  Time of maximum concentration (Tmax) of QRL-101
Pharmacokinetics (plasma): Concentration of QRL-101 before the next dose | Baseline through Follow up Day 5
  Concentration of QRL-101 reached by a drug immediately before the next dose
Pharmacokinetics (plasma): Terminal elimination half-life of QRL-101 | Baseline through Follow up Day 5
  Terminal elimination half-life of QRL-101

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, Principal Investigator — ICON plc
Locations (1):
- ICON plc. Van Swietenlaan 6, Groningen, Netherlands